CLINICAL TRIAL: NCT02949869
Title: Variability of Infant LP Insertion Site Based On Procedural Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Vieira, MD, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00023833
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Traumatic Lumbar Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infant Lumbar Punctures (Experimental): Infants will all be assigned to received two sets of skin markings and sonography exam to assess lumbar puncture landmarks and anatomy.
  Interventions: Other: Spinal Sonography

INTERVENTIONS:
Other: Spinal Sonography — As described previously

SUMMARY:
The reported rate of unsuccessful traditional LP in children (defined as the inability to obtain cerebrospinal fluid or obtaining a traumatic puncture) is as high as 50%. Many factors affect LP success including provider experience. CSF is obtained by puncturing the subarachnoid space (traditionally at the L3-L4 or L4-L5 interspinous process space), and many have hypothesized that the width of this space may predict success. Anecdotally, trainees and those with less experience, tend to perform the LP too low (caudally), where the subarachnoid space tapers, or too laterally (off the midline) resulting in higher failure rates. The investigators seek to determine if planned LP insertion sites vary between training and attendings, and if so, could the decreased success be explained by smaller subarachnoid spaces.

ELIGIBILITY:
Inclusion Criteria:

1. Less than or equal to 12 months of age
2. Availability of a study sonographer to perform bedside ultrasound

Exclusion Criteria:

1. Prior history of LP in preceding 72 hours
2. Known spinal cord abnormality (i.e., tethered cord, spina bifida)
3. Clinically unstable patients (acuity level 1)

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Proportion of Trainee & Attending LP Insertion Sites that are the same | 18 months
  Plan to visualize marked spaces with US to delineate if the trainee and attending marked the same or different interspace (we will quanity the proportion of same interspaces marked and for those that are different, we will quantify the proportion above or below the attending marking)

SECONDARY OUTCOMES:
Subarachnoid Space Width | 18 months
  Measure subarachnoid space width (mm)
Subarachnoid Space Area | 18 months
  Measure subarachnoid space area (mm2)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Vieira, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schreiner RL, Kleiman MB. Incidence and effect of traumatic lumbar puncture in the neonate. Dev Med Child Neurol. 1979 Aug;21(4):483-7. doi: 10.1111/j.1469-8749.1979.tb01652.x. PMID 520695
- [Background] Pinheiro JM, Furdon S, Ochoa LF. Role of local anesthesia during lumbar puncture in neonates. Pediatrics. 1993 Feb;91(2):379-82. PMID 8424014